CLINICAL TRIAL: NCT01725321
Title: Colonoscopy With Narrow Band Imaging for Diagnosis of Proximal Serrated Polyps
Brief Title: Narrow Band Imaging for Diagnosis of Proximal Serrated Polyps
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEUNG Wai Keung, Clinical Professor, The University of Hong Kong
Other Study IDs: NBI_1
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Colonic Neoplasm
Keywords: Colonoscopy; colonic adenoma; serrated polyps
MeSH Terms: conditions — Colonic Neoplasms | interventions — Narrow Band Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Narrow band imaging: Colonoscopy with new narrow band imaging
  Interventions: Other: Narrow band imaging

INTERVENTIONS:
Other: Narrow band imaging — Colonoscopy with new narrow band imaging

SUMMARY:
Although colonoscopy is considered the gold standard for diagnosis of colonic polyps, the missed rate for colonic adenoma ranged from 15-32%. In particular, missed colonic polyps in the right side colon have been suggested to be the cause for interval cancer that developed after a prior negative colonoscopy.

Different endoscopic image enhanced modules like the narrow band imaging (NBI) have been developed to improve colonic polyp detection. However, it remains controversial whether the previous version of NBI helps to improve colonic polyp detection. The new generation colonoscope is equipped with high definition and improved narrow band imaging (NBI) which gives at least twice the viewable distance and contrast. The images obtained are far brighter with better resolution than the previous version. It however remains to be determined whether this enhanced imaging technique could help to improve colonic polyps detection.

Hypothesis:

The new generation NBI increases the detection rate of proximal serrated polyps and reduces the missed rate of all colorectal polyps.

Aims:

* To determine whether the new generation NBI improve the detection rate of proximal serrated polyps.
* To determine whether the new generation NBI improve the detection rate of all colorectal adenoma and polyps.
* To determine whether the new generation NBI reduce the miss rate of colorectal adenoma and polyps.

DETAILED DESCRIPTION:
Design:

Prospective randomized trial

Inclusion:

• All patients scheduled to have screening or scheduled colonoscopy

Exclusion:

* History of Crohn's or ulcerative colitis
* Surveillance for known polyposis syndrome (FAP or HNPCC)
* Previous colonic resection (except appendectomy)
* Refused consent
* Deranged coagulation profile that preclude polypectomy

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to have colonoscopy

Exclusion Criteria:

* History of Crohn's or ulcerative colitis
* Surveillance for known polyposis syndrome (FAP or HNPCC)
* Previous colonic resection (except appendectomy)
* Refused consent
* Deranged coagulation profile that preclude polypectomy

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to have colonoscopy for screening, surveillance or symptoms
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Detection rate of proximal serrated polyp | During colonoscopy
  No. of patients with proximal serrated polyps

SECONDARY OUTCOMES:
Missed rate for proximal serrated polyps | During colonoscopy
  Missing rate for proximal serrated polyps

OTHER OUTCOMES:
Adenoma detection rate | during colonoscopy
  No. of patients with adenoma detected

CONTACTS AND LOCATIONS:
Overall Officials: Wai Keung Leung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China